CLINICAL TRIAL: NCT04033731
Title: Assessment of Stability of Behavioral and Neural Measures of Attention Networks Across Multiple Sessions
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600188; 0217BBRC-02 (Other Grant/Funding Number: *NF/SGVHS Malcom Randall VA Medical Cent)
Record Dates: First submitted 2019-07-19; First posted 2019-07-26 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Stability of Attentional Networks Over Multiple Sessions of Computerized Task
Keywords: cognitive process; visuospatial attention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Controls: Participants will include 15 healthy men and women aged 18-40 years, right-hand dominant, Native English speakers, with normal or corrected-to-normal vision.
  Interventions: Behavioral: Attention Network Task

INTERVENTIONS:
Behavioral: Attention Network Task — The Attention Network Test (ANT) is a computerized cognitive task designed to efficiently probe three independent but interactive attentional networks (alerting, orienting, executive control) in a single task paradigm.
  Other Names: Electroencephalography

SUMMARY:
The purpose of this research study is to learn more about the stability over multiple recording sessions of brainwave activity during a computerized task that measures different types of attention.

DETAILED DESCRIPTION:
Attention is the backbone of cognitive systems and is requisite for other cognitive processes vital to everyday functioning, such as memory, problem solving, language skills, and the cognitive control of behavior. Impairments in attention can result from a variety of factors, such as brain injury, and neurodegenerative and neurodevelopmental disorders, as well as various psychopathologies. A prominent multi-component model of visuospatial attention developed by Posner and colleagues conceptualizes visuospatial attention as an "organ system" comprised of three independent, yet interactive networks which include: 1) Alerting, the generation and maintenance of a vigilant state that facilitates the processing of an upcoming stimulus, 2) Orienting, the disengagement, shifting, and reallocation of attention to a spatial location, and 3) Executive control, the resolution of conflict among competing mutually-exclusive responses that enables selective focus. To aid in understanding of attention, the Attention Network Test (ANT) was developed as a brief computerized measure of the efficiency of each of these networks and has been extensively used in a variety of healthy and clinical populations. Several studies have examined differences in ERPs during the ANT in healthy aging and clinical populations such as ADHD, schizophrenia, and traumatic brain injury (TBI) but have not conducted repeated sessions of the task to evaluate changes over time. While the ANT has been shown to be robustly sensitive to a range of cognitive and/or neuropsychological disorders, the reliability of the ANT across multiple sessions, particularly in terms of neural activity measures, has not been previously examined. An important focus of the proposed research regards the stability of neural measures reflecting activity of each of three different attention networks. One method for examining neural activity involves time locked electroencephalographic (EEG) recordings of brain activity or scalp-recorded brain event-related potentials (ERPs). ERPs can provide insights into the neural correlates of cognitive processes elicited by an experimental task as well as the neural time course. Particularly relevant to this study, the visual N1, a negative-going ERP deflection occurring ~150-200 milliseconds (ms) post-stimulus. N1 amplitude is considered to index attentional allocation. Additionally, a later-occurring positive-going deflection occurring ~300-ms post-stimulus, P3, reflects processes associated with stimulus evaluation and categorization. Previous research in our lab has shown that N1 and P3 are differentially sensitive to attention network functioning probed using the ANT in neurologically-healthy controls and are sensitive to attentional impairment in TBI survivors. Thus, the study team will focus on the stability of N1 and P3 waveforms across the 4 sessions. Previous studies have examined reliability and stability of behavioral measures of the ANT by evaluating the reliability of reaction time (RT) and error rates over multiple sessions. Ishigami reported good temporal stability of network scores across 10 sessions, although some practice effects were seen in orienting and executive-control attention networks. Importantly, no prior work has examined the temporal stability of ERPs with repeated ANT performance, which is among the primary aims of the proposed research. Finally, in an exploratory manner, the investigators will extend findings from one of our earlier studies demonstrating altitudinal attentional biases for upper vertical space in healthy participants and the absence of such biases in TBI survivors. Specifically, the investigators will examine which of three attentional networks are sensitive to such biases in healthy controls and determine the ERP signatures of these biases.

ELIGIBILITY:
Inclusion Criteria:

* right-hand dominant
* Native English speakers
* with normal or corrected-to-normal vision

Exclusion Criteria:

* Not right-hand dominant
* Does not speak english as a native language
* No history of neurological disorder such as stroke, epilepsy or chronic seizure disorder, traumatic brain injury or concussion, psychiatric disorder such as schizophrenia, bipolar disorder, major depression or anxiety disorder, any psychiatric inpatient hospitalization for any of these disorders, or previously diagnosed learning disability
* Currently taking any prescribed medications for anxiety, depression, or seizures
* Alcohol use more than 3 days a week

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Controls
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Change in the temporal stability of behavioral measures of three attention networks: change in reaction time across four sessions | Week 1; Week 2; Week 3; Week 4
  The Attention Network Task (ANT) combines a covert cuing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention. These distinct components of attention are: alerting, orienting, and executive control. These facets of attention will be assessed at 4 time points scheduled 1 week apart as follows: ANT Alerting Reaction Time score, ANT Orienting Reaction Time score and ANT Executive-control Reaction Time score. The lower the score the faster the reaction time.
Change in the temporal stability of neural measures of three attention networks using scalp-recorded electroencephalography (EEG) | Week 1; Week 2; Week 3; Week 4
  Scalp-recorded brain event related potentials (ERP) will be acquired from 64 EEG sensors while participants perform the ANT reflecting alerting, orienting, and executive control components of attention. These facets of attention will be assessed at 4 time points scheduled 1 week apart. ANT alerting will be interrogated by examining the amplitude of the P300 component of the ERP in microvolts, as will orienting and executive-control.

CONTACTS AND LOCATIONS:
Overall Officials: William Perlstein, PhD, Principal Investigator — University of Florida
Locations (1):
- College of Public Health and Health Professions, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No